CLINICAL TRIAL: NCT04087408
Title: Role of Triptorelin 0.1 mg as a Luteal Phase Support in Assisted Reproductive Technique After Embryo Transfer : a Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moustafa Mohammed Abouelea (Other)
Responsible Party: Sponsor-Investigator, Moustafa Mohammed Abouelea, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MMAbouelea
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Effect of Adding GnRHa as Luteal Phase Support in Antagonist ART Cycles
Keywords: GnRHa , LPD, antagonist, progesterone and ART

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): 1. Ovarian stimulation will be initiated from the day 2 of the menstrual cycle using gonadotropins 150-450 IU
  2. doses will be adjusted according to ovarian response. Once the leading follicle will reach a size of 14 mm, co-treatment with a GnRH antagonist will initiated and continued up until at least three follicles reached a size of 17-18 mm.
  3. Trigger will be done using HCG followed by OPU 36 h later.
  4. Retrieved oocytes will be fertilized by ICSI.
  5. LPS, using micronized P (400 mg/day) vaginally beginning on the day of oocyte retrieval.
  6 - Blood sampling will be performed for progesterone 7 days after OPU.
  7-Quantative BHCG will be performed 14 days after OPU.
- study group (Active Comparator): 1. Ovarian stimulation will be initiated from the day 2 of the menstrual cycle using gonadotropins 150-450 IU
  2. doses will be adjusted according to ovarian response. Once the leading follicle will reach a size of 14 mm, co-treatment with a GnRH antagonist will initiated and continued up until at least three follicles reached a size of 17-18 mm.
  3. Trigger will be done using HCG followed by OPU 36 h later.
  4. Retrieved oocytes will be fertilized by ICSI.
  5. LPS, using micronized P (400 mg/day) vaginally beginning on the day of oocyte retrieval.
  6. GnRH agonist 0.1 mg will be given 6 days after OPU.
  7. Blood sampling will be performed for progesterone within 24 h following the GnRH agonist 0.1 mg
  8. Quantative BHCG will be performed 14 days after OPU.
  Interventions: Drug: Effect of adding gonadotropins releasing hormone agonist to progesterone for luteal phase support in assisted reproductive technique )antagonist cycles(: a randomized controlled trial

INTERVENTIONS:
Drug: Effect of adding gonadotropins releasing hormone agonist to progesterone for luteal phase support in assisted reproductive technique )antagonist cycles(: a randomized controlled trial — 1. Ovarian stimulation will be initiated from the day 2 of the menstrual cycle using gonadotropins 150-450 IU
  2. doses will be adjusted according to ovarian response. Once the leading follicle will reach a size of 14 mm, co-treatment with a GnRH antagonist will initiated and continued up until at least three follicles reached a size of 17-18 mm.
  3. Trigger will be done using HCG followed by OPU 36 h later.
  4. Retrieved oocytes will be fertilized by ICSI.
  5. LPS, using micronized P (400 mg/day) vaginally beginning on the day of oocyte retrieval.
  6. GnRH agonist 0.1 mg will be given 6 days after OPU for the study group.
  7. Blood sampling will be performed for progesterone within 24 h following the GnRH agonist 0.1 mg
  8. Quantative BHCG will be performed 14 days after OPU.
  Arms: study group

SUMMARY:
There is still controversy over the best LPS agent and protocol and its dose and duration as well as the time of initiation and cessation.

There are many protocols of luteal support in assisted reproductive technology (ART) cycles. Luteal phase support with progesterone is a standard approach for ART cycles .

Initial studies in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) patients have demonstrated that the use of a GnRH agonist (GnRHa) trigger, followed by fresh transfer and a standard luteal phase support (LPS) was associated with unacceptably high rates of loss in early pregnancy compared to hCG trigger, particularly in normal responder (NR) patients.

During IVF and fresh embryo transfer, the luteal function is disrupted and the success of the treatment is critically dependent on exogenous luteal phase support

During the last decade, two different modified LPS strategies have been proposed to overcome the mentioned luteal phase deficiency. One of these approaches has been called the "European approach" in which the endogenous steroid (progesterone and estradiol) production by the corpora lutea is boosted by exogenous LH activity, i.e., LH or hCG after GnRHa trigger. The other approach has been called the "American approach" in which luteal progesterone and estradiol are administered exogenously, thus, disregarding the function of the corpora lutea.

It has been subsequently concluded that this early pregnancy loss was caused by luteal phase (LP) insufficiency, despite the use of a standard LPS package of progesterone (P) and estradiol (E2). The LP defect was primarily caused by reduced early-mid-luteal luteinizing hormone (LH) activity, resulting in a significant reduction in progesterone output by the corpora lutea (CL) as no adverse effects were seen with respect to the maturity rate of oocytes, fertilization rates, embryo quality, and reproductive outcomes during the subsequent replacement of frozen embryos derived from women who had received a GnRHa trigger .

Transvaginal progesterone is commonly used for luteal phase support. Progesterone administration is initiated on the oocyte pick-up (OPU) day and continued for 12 days, until the serum beta human chorionic gonadotropin (hCG) measurement day. However, there are conflicting results regarding the dose, route of administration (oral, subcutaneous, transvaginal), duration (until the ultrasound demonstration of heartbeat in an intrauterine gestational sac, until 10 weeks of gestation, until 12 weeks of gestation), and formulations such as synthetic or micronized types of progesterone.

A bolus of GnRHa, when administered 6 days after OPU in GnRH antagonist cycles, is able to induce a surge of pituitary gonadotropins (FSH and LH), eliciting an increase in steroid production (E2 and P) by the CL.

The exact mechanism behind the presumed beneficial effect of LP GnRHa administration remains poorly defined. It has been hypothesized that GnRHa either supports CL function by inducing LH secretion by the pituitary gonadotrophic cells or stimulates the endometrial GnRH receptors.

Tesarik postulated a direct effect of GnRHa on the embryo, as suggested by an increase in β-HCG secretion.

Importantly, there are significant differences in the early-mid-LP endocrine pattern when GnRHa triggers and hCG triggers are compared, especially in terms of LH levels. From this, it could be hypothesized that the GnRHa-triggered IVF cycle could benefit more from the addition of a bolus of GnRHa to boost the circulating endogenous LH and thus, progesterone levels around the time of implantation than the hCG triggered cycle. No studies previously investigated this issue. Therefore, the aim here was to explore a possible fine-tuning of the LPS of GnRHa-triggered IVF/ICSI cycles, using the previously suggested protocol.

Significantly increased implantation rates (IRs) were previously reported in oocyte recipients as well as in patients who were triggered with hCG, if they received a single mid-luteal bolus of GnRHa in addition to standard LPS .

A beneficial effect of a single dose of GnRH agonist administration as a luteal phase supporting agent is yet to be determined because of the wide heterogeneity of data present in literature. Well-designed randomized clinical studies are required to clarify any effect of luteal GnRH agonist addition on pregnancy outcome measures with different doses, timing, and administration routes of GnRH agonists .

Administration of 0.1 mg of the GnRH agonist triptorelin on day 3 after embryo transfer led to a significant improvement in implantation rate (12.3% vs. 7.3%) and clinical pregnancy rate (25.5% vs. 10.0%) as compared with placebo.

Luteal phase support with single-dose GnRHa might be as efficient as three doses of hCG. Large prospective, randomized-controlled studies are required comparing GnRHa and hCG for luteal phase support.

DETAILED DESCRIPTION:
Type of the study: Open labelled randomized controlled trial

Study Setting: ART Unit, Women's Health Hospital

c. Sample Size Calculation: Sample size calculation was calculated using Epi Info software (version 7). Based on previous study the pregnancy rate was 32.6% with GnRHa and 12.5% with control. Based on these percentages and with a confidence level of 95% and power of 80%, the sample size needed for the study was estimated to be 150 women (75 in each group).

Study tools :

All women scheduled for ICSI cycles in the AUH -ART unit and fulfil the above criteria will be invited to participate in the study, and subjected to the following

1. A Thorough history will be taken with special emphasis on age and parity of the patients, age and duration of marriage, menstrual pattern, contraceptive history (with stress on type and duration of use), type and duration of infertility and type of previous delivery.
2. Blood sampling will be performed for baseline evaluation FSH, LH, TSH and AMH on 2nd day of menses.
3. Ovarian stimulation will be initiated from the day 2 of the menstrual cycle using recombinant gonadotropins 150-450 IU depending on patient age, BMI, antral follicle count and basal serum FSH.
4. After 5 days, doses will be adjusted according to ovarian response. Once the leading follicle will reach a size of 14 mm, co-treatment with a GnRH antagonist will initiated and continued up until at least three follicles reached a size of 17-18 mm.
5. Trigger will be done using HCG followed by OPU 36 h later.
6. Retrieved oocytes will be fertilized by ICSI depending on sperm quality.
7. According to the local regional policy and after an agreement between the patient and the medical team, one to three embryos will be transferred.
8. For LPS, all patients will receive micronized P (400 mg/day) vaginally beginning on the day of oocyte retrieval and continuing until either end of first trimester by ultrasound or a negative pregnancy test.
9. For the study group GnRH agonist 0.1 mg will be given 6 days after OPU.
10. Blood sampling will be performed for progesterone within 24 h following the GnRH agonist 0.1 mg injection particularly in the study group.
11. Blood sampling will be performed 14 days after OPU for Quantative BHCG.

Randomization:

Randomization will be accomplished by using cards at the time of embryo transfer; two hundred will sequentially divide into two groups. Opaque sealed envelopes will used containing 75 cards labelled control group and 75 cards labelled study group. All of envelops will mixed together randomly in a box. The cards will be pulled randomly.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 40 years.
2. Baseline FSH > 10 IU/L.
3. Fresh stimulated cycles
4. Antagonist cycles

Exclusion Criteria:

1. Uterine fibroid if encroaching uterine cavity.
2. Mullerian anomalies.
3. Ovarian endometrioma.
4. Adnexal hydrosalpinx "except after disconnection".
5. Ovarian hyper stimulation syndrome (OHSS) an exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations. It is classified as mild, moderate, or severe according to the degree of abdominal distention, ovarian enlargement, and respiratory, hemodynamic and metabolic complications.
6. Poor responders according to bologna criteria.
7. Women refused to participate in an RCT.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 1. Age between 20 to 40 years.
  2. Baseline FSH > 10 IU/L.
  3. Fresh stimulated cycles
  4. Antagonist cycles
Enrollment: 150 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing clinical pregnancy rate | up to 7 weeks pregnancy
  the number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles, or embryo transfer cycles

SECONDARY OUTCOMES:
Implantation rate. | up to 4 weeks of pregnancy
  implantation rate "the number of gestational sacs observed divided by the number of embryos transferred"
First trimester abortion | up to 13 weeks of pregnancy
  abortion before 12 weeks of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt